CLINICAL TRIAL: NCT01190072
Title: LIPID-LOWERING THERAPY FOR SECONDARY PREVENTION IN PATIENTS UNDERGOING ELECTIVE PERCUTANEOUS CORONARY INTERVENTION (PCI) A 10-week, Open-label, Non-interventional Study of Total Cholesterol/LDL-cholesterol Management in Real Life in Coronary Patients Hospitalised for Elective PCI
Brief Title: Lipid-lowering Therapy for Secondary Prevention in Patients Undergoing Elective Percutaneous Coronary Intervention (PCI)
Status: Terminated | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CSI-DUM-2010/1
Record Dates: First submitted 2010-08-26; First posted 2010-08-27 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Coronary Artery Disease
Keywords: Blood lipids; percutaneous coronary intervention; lipid lowering treatment
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to follow the management of blood lipids in patients with planned percutaneous coronary intervention (widening of coronary vessels) in a period from 6 to 10 weeks after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Male or nonpregnant female
* Coronary patient hospitalised for elective PCI
* Hypercholesterolaemia defined as LDL-C ≥ 2 mmol/L

Exclusion Criteria:

* Any chronic inflammatory condition
* Chronic anti-inflammatory pharmacotherapy (except low-dose ASA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Secondary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2010-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Serum total cholesterol concentration | Week 0
Serum total cholesterol concentration | Once during the time period between Week 6 and Week 10
Serum LDL cholesterol concentration | Week 0
Serum LDL cholesterol concentration | Once during the time period between Week 6 and Week 10

SECONDARY OUTCOMES:
Proportion of patients achieving LDL-C < 2 mmol/L | Once during the time period between Week 6 and Week 10
Proportion of patients achieving total cholesterol < 4 mmol/L | Once during the time period between Week 6 and Week 10
Change of hsCRP levels from baseline | Once during the time period between Week 6 and Week 10

CONTACTS AND LOCATIONS:
Overall Officials: Vojko Kanic, Principal Investigator — University Medical Centre Maribor
Locations (1):
- Research Site, Maribor, Slovenia